CLINICAL TRIAL: NCT00509444
Title: Cancer Prevention and Treatment Among African American Older Adults
Brief Title: Cancer Prevention and Treatment Among African American Older Adults: Treatment Trial
Acronym: CPTD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jean Ford, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Colon Cancer; Rectum Cancer; Cervix Cancer; Prostate Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Uterine Cervical Neoplasms; Prostatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational materials (Active Comparator)
  Interventions: Behavioral: Educational materials
- Educational materials, plus patient navigation (Experimental)
  Interventions: Behavioral: educational materials, plus patient navigation

INTERVENTIONS:
Behavioral: Educational materials
  Arms: Educational materials
Behavioral: educational materials, plus patient navigation
  Arms: Educational materials, plus patient navigation

SUMMARY:
The Centers for Medicare and Medicaid Services (CMS) has awarded cooperative agreements to 6 sites from across the country (Salt Lake City, UT, Molokai, HI, Houston, TX, Newark, NJ, Detroit, MI, and Baltimore City) to participate in a national 4-year demonstration (September 15, 2006 to September 30, 2010). One goal of the demonstration is to reduce disparities in cancer treatment among seniors from U.S. racial and ethnic minority populations. Each site will focus on a specific racial/ethnic minority group, and collaborate with CMS in project implementation. A Core questionnaire, the Cancer Screening Assessment (CSA) will be administered at baseline to all participants in the demonstration. Participant identification, randomization, and intervention implementation will be standardized across sites.

Goal: The proposal developed by the Johns Hopkins Bloomberg School of Public Health in collaboration with the Baltimore City Community Health Coalition is designed to address persistent disparities in breast, cervix, colon/rectum, prostate and lung cancer treatment.

Primary Objective: Conduct A CONTROL RANDOMIZED TRIAL within a randomized control demonstration project (N = 200) to compare the efficacy of 2 interventions that differ in intensity to improve continuity and outcomes of care among African Americans seniors. Among African American seniors, compared to a less intensive intervention (general information and educational materials), does the addition of facilitation services delivered by a health coordinator result in a greater improvement in adherence to recommended treatment among those diagnosed with breast, cervix, colon/rectum, prostate, or lung cancer?

Study Population: We will recruit African Americans, age 65 years or older, and currently enrolled in Medicare Parts A and B. (Baltimore City's 82,202 seniors represent 13% of its population, and account for 68% of the City's cancer deaths. Among these seniors, 96% have Medicare Parts A and B, 54.5% have income levels at less than 250% of the federal poverty guideline, and 55.6% are African American.)

The trial consists of individuals diagnosed with breast, cervical, colorectal, prostate, or lung cancer. Eligible participants will respond to a baseline questionnaire, the Cancer Screening Assessment (CSA). They will then be randomized to receive a less intensive or more intensive intervention. The less intensive group will receive general information about cancer and Medicare covered services and instructions to discuss the information with their primary care doctor. The more intensive group will receive the same information as the less intensive group receives, plus tailored facilitation services delivered by a nurse-supervised community health worker. The primary outcome variable for the trial will be the difference between randomized groups in adherence to treatment for breast, cervix, colon/rectum, prostate and lung cancer.

A community advisory committee will guide all aspects of the study and will include important stake holders (both public and private sectors), representatives from the Baltimore City Community Health Coalition, the Baltimore City Department of Health, the Maryland Department of Health and Mental Hygiene, community leaders, consumers, health care providers (physicians, oncologists, nurse practitioners, physician assistants, nurses, social workers, pathologists) and academicians.

DETAILED DESCRIPTION:
Among African American seniors, compared to a less intensive intervention (general information and educational materials), does the addition of facilitation services delivered by a health coordinator result in a greater improvement in adherence to recommended treatment among those diagnosed with breast, cervix, colon/rectum, prostate, or lung cancer?

Background The Centers for Medicare and Medicaid Services (CMS) received congressional authorization to launch a nationwide demonstration project to address persistent disparities in cancer treatment among racial and ethnic minority populations. Hopkins was selected as one of six national sites to conduct a demonstration project designed to test an intervention strategy to promote adherence to cancer treatment.

Aim This demonstration project will evaluate the efficacy of a health coordinator model. We will conduct A RANDOMIZED CONTROLLED TRIAL testing the efficacy of the intervention for African American seniors diagnosed with cancer. The duration of follow-up post-randomization will be from date of randomization and September 30th, 2010, the end date for the demonstration.

This randomized controlled trial will compare the efficacy of a less intensive intervention (general information and educational materials in the context of "usual care") to that of a more intensive intervention, the addition of a health coordinator (HC), in promoting adherence to treatment among African American seniors who have been diagnosed with breast, cervix, colon/rectum, prostate or lung cancer.

The primary outcome variable for the trial will be the difference between the two intervention groups in the time to initiation of therapy, beginning on the date of randomization.

Population: The study population will consist of a convenience sample of 200 individuals diagnosed with breast, cervix, colon, lung or prostate cancer, and who intend to receive their cancer treatment from either Johns Hopkins Hospital (JHH) or from Johns Hopkins Bayview Medical Center (JHBMC).

The sampling frame will be restricted to African American Medicare beneficiaries, age 65 and older, enrolled in Medicare Parts A and B, but not enrolled in managed care (Medicare Part C), hospice, or some other extended care facility. With a population of 651,154, African Americans constitute 64% of Baltimore City's total population44. Additionally, 13.2% of Baltimoreans are age 65 or older, and this accounts for 68% of the City's cancer deaths.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Enrolled in Medicare Part A
* Enrolled in Medicare Part B of Title XVIII of the Social Security Act
* Provided Informed Consent
* Diagnosed with breast, cervical, colorectal, prostate, or lung cancer AND 1) have not yet begun treatment for this cancer; or 2) are currently receiving treatment or received a last treatment within the past five years; or 3) received a last treatment 5 or more years ago but have been in remission less than 5 years; AND 4) intend to receive cancer treatment from either Johns Hopkins Hospital (JHH) or from Johns Hopkins Bayview Medical Center (JHBMC)

Exclusion Criteria:

* Age less than 65
* Enrollment in Medicare managed care (Part C)
* Residence in a chronic care facility or otherwise institutionalized
* Planning to move within the next year
* Unable or unwilling to give informed consent
* Another member of the household enrolled in the demonstration project
* Diagnosed with breast, cervical, colorectal, prostate, or lung cancer and received a last treatment for this cancer 5 or more years ago and have been in remission for 5 or more years
* Currently receiving treatment or will be receiving treatment soon for a non-study cancer
* Currently diagnosed with a non-study cancer and have not received treatment yet for this cancer but returning for additional tests and observation
* Diagnosed with a non-study cancer and received the last treatment within the last 5 years
* Diagnosed with a non-study cancer and received the last treatment for this cancer 5 or more years ago and have been in remission less than 5 years
* Diagnosed with a non-study cancer and received the last treatment for this cancer 5 or more years ago and have been in remission for 5 or more years
* Diagnosed with a study cancer and being treated outside of Johns Hopkins Medical Institutions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be difference between the two intervention groups in the time to initiation of therapy, beginning on the date of randomization.

SECONDARY OUTCOMES:
The time in days to the first treatment-related visit (with a medical, radiation oncologist, or surgical oncologist) beginning on the date of randomization.
The rate of completion of recommended courses of chemo and/or radiation therapy.
The proportion completing recommended surgical treatment.
The proportion receiving recommended screenings for breast, cervix, colon/rectum and prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jean G. Ford, MD, Principal Investigator — Bloomberg School of Public Health, Baltimore, Maryland, United States
Locations (1):
- Bloomberg School of Public Health, Baltimore, Maryland, United States